CLINICAL TRIAL: NCT04942652
Title: An Open-label, Three-period, One-sequence Crossover Clinical Trial to Evaluate the Effects of Food or Proton Pump Inhibitor on the Pharmacokinetics of Itraconazole in Healthy Volunteers
Brief Title: Study to Evaluate Effects of Food or Proton Pump Inhibitor on the Pharmacokinetics of Itraconazole in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeungHwan Lee, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Itraconazole_pH
Record Dates: First submitted 2021-06-20; First posted 2021-06-28 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Achlorhydria
MeSH Terms: conditions — Achlorhydria | interventions — Itraconazole; Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Itraconazole 200 mg under fasted condition (Experimental): A single oral administration of itraconazole 200 mg under fasted condition
  Interventions: Drug: Itraconazole 200 mg
- Itraconazole 200 mg under fed condition (Experimental): A single oral administration of itraconazole 200 mg under fed condition
  Interventions: Drug: Itraconazole 200 mg
- Esomeprazole 40 mg + Itraconazole 200 mg under fasted condition (Experimental): Oral administration of esomeprazole 40 mg once daily for 6 days and then a single oral administration of itraconazole 200 mg under fasted condition
  Interventions: Drug: Itraconazole 200 mg; Drug: Esomeprazole 40 mg

INTERVENTIONS:
Drug: Itraconazole 200 mg — Itraconazole 100 mg capsule x 2
  Other Names: Sporanox capsule
Drug: Esomeprazole 40 mg — Esomeprazole 40 mg tablet x 1
  Other Names: Nexium
  Arms: Esomeprazole 40 mg + Itraconazole 200 mg under fasted condition

SUMMARY:
The aim of this study is to evaluate the effects of food or proton pump inhibitor on the pharmacokinetics of itraconazole in healthy volunteers.

DETAILED DESCRIPTION:
Evaluation criteria

* Pharmacokinetic assessment with plasma concentrations of itraconazole and hydroxy-itraconazole
* Safety assessments with adverse event monitoring including subjective/objective symptoms, physical examination, vital signs, and laboratory tests

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged ≥ 19 years and ≤ 50 years at the time of screening
* Body weight of ≥ 55.0 kg and ≤ 90.0 kg, with body mass index (BMI) of ≥ 19.0 kg/m2 and ≤ 30.0 kg/m2 at the time of screening
* A subject without any congenital or chronic disease, and has no medical examination result as pathological symptoms or signs
* A subject who listened to sufficient explanation and fully understood this study, and voluntarily decided to participate and agreed in writing to comply with the precautions
* A subject determined eligible for this study by investigator based physical examination, clinical laboratory tests, interview, etc.

Exclusion Criteria:

* A subject with clinically significant hepatobiliary (severe hepatic impairment, etc.), renal (severe renal impairment, etc.), neurologic, immunologic, respiratory, gastrointestinal, endocrine, blood•oncology, cardiovascular (heart failure, Torsades de pointes, etc.), urinary, or, psychical diseases (except for simple dental past history such as tartar, impacted tooth, or wisdom tooth) or a history
* A subject who has hypersensitivity to the investigational products, drugs containing the same class, or other drugs (penicillin and antibiotics, etc.), or a history of clinically significant hypersensitivity
* A subject with a history of gastrointestinal disorders (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux disease, Crohn's disease, etc.) or surgery (except for simple appendectomy and herniotomy) that may affect the safety and pharmacokinetics of the investigational products
* A subject with the following results in the screening test:

  1. Blood AST (GOT), ALT (GPT): > Normal range upper × 1.5
  2. QTc interval: > 450 ms
  3. Positive serological test (syphilis test, hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test)
* A subject with systolic blood pressure < 80 mmHg or > 160 mmHg, or diastolic blood pressure < 50 mmHg or > 100 mmHg when vital signs are measured in sitting position after resting for at least 3 minutes
* A subject with a history of drug abuse
* A subject who administered any prescription drugs or herbal medicine within 2 weeks prior to the expected date of the first dose, or any over-the-counter drug (OTC drug, health functional food or vitamin within 1 week prior to the expected date of the first dose (However, can participate in the study if otherwise decided eligible by the investigator), or is expected to administer it
* A subject who administered drugs that induce (such as barbitals) or inhibit (such as clarithromycin) the drug metabolizing enzymes within 1 month prior to the expected date of the first dose
* A subject who participated in other clinical trial or bioequivalence study within 6 months prior to the expected date of the first dose
* A subject who donated whole blood within 2 months or the component blood within 1 month prior to the expected date of the first dose, or received blood transfusion within 1 month prior to the expected date of the first dose
* A subject with persistent alcohol intake (> 21 units/week, 1 unit = 10 g of pure alcohol), or inability to abstain from drinking from 3 days before the expected date of the first dose until the last discharge
* A subject with inability to refrain from grapefruit-containing food from 3 days before the expected date of the first dose until the last discharge
* A subject with excessive caffeine intake (> 5 units/day), or inability to refrain from caffeine or caffeine-containing food from 3 days before the expected date of the first dose until the last discharge
* A subject with inability to use a medically acceptable double contraception or contraception throughout the study and for at least 4 weeks after the last dose, and with inability to agree to donate sperm until the period

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Cmax of itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of itraconazole
AUClast of itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of itraconazole
AUCinf of itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of itraconazole
Tmax of itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of itraconazole
t1/2 of itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of itraconazole
CL/F of itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of itraconazole
Vd/F of itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of itraconazole
Cmax of hydroxy-itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of hydroxy-itraconazole
AUClast of hydroxy-itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of hydroxy-itraconazole
AUCinf of hydroxy-itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of hydroxy-itraconazole
Tmax of hydroxy-itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of hydroxy-itraconazole
t1/2 of hydroxy-itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of hydroxy-itraconazole
metabolic ratio of hydroxy-itraconazole | Day 1/Day 8/Day 16 pre-dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 hour post-dose
  Pharmacokinetic parameters of hydroxy-itraconazole

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided